CLINICAL TRIAL: NCT03882736
Title: Prospective Study of Volumetric Gluteal Region by Parasacral Perforator Flaps in Circumferential Body Lift
Brief Title: Volumetric Study of the Buttocks After Flap Augmentation in Buttocks Lifting
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0036
Record Dates: First submitted 2019-01-24; First posted 2019-03-20 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Weight Loss
Keywords: plastic and reconstructive surgery; gluteal ptosis; platipygia
MeSH Terms: conditions — Weight Loss | interventions — Surgical Flaps; Body Contouring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: gluteal augmentation with flap in circumferential body lift — classic circumferential bodylift surgery, using two different well-known flaps for gluteal augmentation

SUMMARY:
The development of bariatric surgery, its effectiveness and the reduction of complications are at the origin of massive weight loss, the corollary of which has been a clear increase in the demands of treatment of sequelae of weight loss.

ELIGIBILITY:
Inclusion criteria:

* 12 months minimum delay with bariatric surgery
* female, BMI<30kg/m2
* Age greater than or equal to 18 years
* Stable weight for more than 6 months
* lack of volume in gluteal region
* agree with clinical trial

Exclusion criteria:

* Patient under tutorship or curatorship
* Pregnancy or breastfeeding
* hemoglobinemia< 12g/dL
* Albuminemia<3,5g/dL
* active smoking more than 1 month before surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients after massiv weight loss who come in toulouse or montpellier hospital to take care of slimming effects
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Volumetric increase by para-sacral flap | day before the operation
  evaluate the gluteal volume after augmentation with a parasacral flap using a 3D camera
Volumetric increase by para-sacral flap | then at the 3th month post surgery
  evaluate the gluteal volume after augmentation with a parasacral flap using a 3D camera
Volumetric increase by para-sacral flap | then at the 6th month post surgery
  evaluate the gluteal volume after augmentation with a parasacral flap using a 3D camera

SECONDARY OUTCOMES:
Clinical evolution | During hospitalization (Day 0 to Day 5)
  Results of clinical evaluation : look for seroma andhematoma during hospitalization
Results of clinical evolution | Day 15
  clinical evaluation : look for seroma and hematoma post surgery
Results of clinical evolution | 2nd week after surgery
  clinical evaluation : look for seroma and hematoma then at the 2nd week after surgery
Results of clinical evolution | 3rd week after surgery
  clinical evaluation : look for seroma and hematoma then at 3rd week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Farid BEKARA, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France